CLINICAL TRIAL: NCT03380975
Title: Role of Montelukast in Asthma and Allergic Rhinitis Patients
Acronym: MAAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinision (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN/PK/MAAP/SP/2017-01
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2017-12

CONDITIONS: Asthma and Allergic Rhinitis
Keywords: MAAP; Asthma; Allergic rhinits
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: Montelukast is an orally active compound which binds with high affinity and selectivity to the CysLT1 receptor. Montelukast inhibits physiologic actions of LTD4 at the CysLT1 receptor without any agonist activity. As a result, bronchoconstriction is inhibited with decreased airway and blood eosinophil's leading to improved control over asthma and allergic rhinitis
Masking Description: Montelukast is an orally active compound which binds with high affinity and selectivity to the CysLT1 receptor.Montelukast should be taken once daily in the evening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Montelukast 10 mg (Experimental): Montelukast is an orally active compound which binds with high affinity and selectivity to the CysLT1 receptor. Montelukast inhibits physiologic actions of LTD4 at the CysLT1 receptor without any agonist activity. As a result, bronchoconstriction is inhibited with decreased airway and blood eosinophil's leading to improved control over asthma and allergic rhinitis.
  Interventions: Drug: Montelukast 10mg

INTERVENTIONS:
Drug: Montelukast 10mg — Montelukast is an orally active compound which binds with high affinity and selectivity to the CysLT1 receptor. Montelukast inhibits physiologic actions of LTD4 at the CysLT1 receptor without any agonist activity. As a result, bronchoconstriction is inhibited with decreased airway and blood eosinophil's leading to improved control over asthma and allergic rhinitis. Montelukast should be taken once daily in the evening
  Other Names: Aireez

SUMMARY:
To determine the effect of Montelukast in Asthma and Allergic rhinits patients

DETAILED DESCRIPTION:
Montelukast is a potent and selective blocker of the CysLT1 receptor. Accordingly, a recent study has shown that Montelukast can improve symptoms of seasonal allergic rhinitis and asthma in patients with both diseases. For treatment of asthma, Montelukast is administered once daily to adults as a 10-mg film-coated tablet, to children aged 6-14 years as a 5-mg chewable tablet, and to children aged 2-5 years as a 4-mg chewable tablet form. Asthma and allergic rhinitis have been linked clinically for many years as "one airway one diseases". Patients with allergic asthma and rhinitis are significantly more likely to experience asthma attacks compared to patients with asthma alone. Side effects most commonly reported above placebo included headache, otitis media, upper respiratory infection, and pharyngitis

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Signed Informed Consent
* Clinical diagnosis of Asthma and Allergic Rhinitis

Exclusion Criteria:

* Previous adverse reaction to Montelukast
* History of hyper-eosinophilic disorder other than atopic disease
* Female subjects who are pregnant, breast-feeding
* Any significant and active pulmonary pathology other than asthma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of montelukast on asthma day and night symptoms changes from baseline after 4 weeks of treatment | 4 weeks
  To determine the efficacy of montelukast on asthma day and night symptoms changes from baseline after 4 weeks of treatment [Designated as safety issue: No] [Time Frame: 0 days to 4 weeks]

SECONDARY OUTCOMES:
Efficacy of montelukast on allergic rhinitis symptoms changes from baseline after 4 weeks of treatment | 4 weeks
  To determine the efficacy of montelukast on allergic rhinitis symptoms changes from baseline after 4 weeks of treatment [Designated as safety issue: No] [Time Frame: 0 days to 4 weeks]
Effect of montelukast in change in individual quality of life using Quality of life questionnaire after 4 weeks of treatment | 4 weeks
  To determine the effect of montelukast in change in individual quality of life using Quality of life questionnaire after 4 weeks of treatment [Designated as safety issue: No] [Time Frame: 0 days to 4 weeks]
Proportion of participants experiencing an adverse event (AE) | 4 weeks
  Proportion of participants experiencing an adverse event (AE) [Designated as safety issue: Yes] [Time Frame: 0 days to 4 weeks]

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Faiyaz, FCPS,FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dr. Faisal Faiyaz Zuberi, Karachi, Sindh, Pakistan